CLINICAL TRIAL: NCT07193784
Title: Effect of Reiki Applied After Coronary Angiography on Pain and Comfort Level: A Randomized Single-blind Placebo-controlled Study
Brief Title: Effect of Reiki Applied After Coronary Angiography on Pain and Comfort Level
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Abdullah Avcı, Abdullah Avcı, PhD, Principal Investigator, Nursing Services Coordinator, Mersin University Hospital, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVCI-MERSİN-2025
Record Dates: First submitted 2025-08-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Coronary Angiography
Keywords: coronary angiography; reiki; pain; comfort
MeSH Terms: conditions — Pain | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, placebo-controlled, parallel-group trial with three arms (Reiki, sham Reiki, and control). Participants are allocated in a 1:1:1 ratio and receive only the intervention assigned to their group. No crossover between arms is planned.
Who Masked: Participant
Masking Description: Participants are blinded to their group allocation. Reiki and sham Reiki sessions are delivered in identical settings (duration, environment, body position, and practitioner interaction) to maintain blinding. Practitioners, who also serve as data collectors, are aware of the intervention type due to the nature of the technique. Statistical analysis will be performed by an independent researcher blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reiki (Experimental): Participants receive a 30-minute Reiki session by a trained practitioner after coronary angiography. Pain and comfort are assessed at four time points.
  Interventions: Behavioral: Reiki
- Sham reiki (Placebo Comparator): Participants receive a 30-minute sham Reiki session mimicking Reiki hand positions without actual energy intervention. Pain and comfort are assessed at the same time points.
  Interventions: Behavioral: Sham reiki
- Control (No Intervention): Participants receive standard post-angiography care without any Reiki or sham intervention. Pain and comfort are assessed at the same time points.

INTERVENTIONS:
Behavioral: Reiki — Reiki therapy applied by trained practitioner for 30 minutes.
  Arms: Reiki
Behavioral: Sham reiki — Sham Reiki applied by same practitioner, mimicking Reiki without actual energy technique.
  Arms: Sham reiki

SUMMARY:
Coronary angiography is an invasive imaging technique that directly visualizes the anatomical structure of the coronary arteries and is considered the gold standard for diagnosing significant coronary artery disease. In the post-coronary angiography period, alleviating pain and enhancing patient comfort are important goals of clinical care. Reiki is an energy-based complementary therapy aimed at supporting the body's natural healing processes and promoting relaxation. Among non-pharmacological interventions, Reiki-a practice rooted in Traditional Chinese Medicine and meaning universal life energy-is a safe, cost-effective, and easily applicable method. Studies have shown that Reiki is effective in reducing pain, anxiety, fear, and stress, as well as in improving comfort and holistic well-being. This study was designed to examine the effects of Reiki therapy administered after coronary angiography on patients' levels of pain and comfort.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years.
* Undergoing coronary angiography for the first time.
* No additional interventions (e.g., stent placement) performed during angiography.
* Coronary angiography performed via femoral artery.
* Elective (non-emergency) coronary angiography.
* No prior experience with Reiki, Therapeutic Touch, or other energy therapies.
* Able to understand and speak Turkish.
* Open to communication and able to participate in face-to-face interviews.

Exclusion Criteria:

* Development of acute complications during or after coronary angiography (e.g., myocardial infarction, severe arrhythmia, embolism, bleeding at the intervention site, hematoma).
* Any diagnosed psychiatric disorder.
* History of chronic pain or regular use of analgesics.
* Previous experience with Reiki or similar complementary therapies.
* Requirement for sedative or opioid analgesic use during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Pain level | Baseline (before intervention), 30 minutes after intervention, 2 hours after intervention, and prior to first mobilization (within 24 hours).
  Pain intensity measured using Visual Analog Scale (VAS, 0-10) via face-to-face interviews at the specified time points.

SECONDARY OUTCOMES:
Comfort level | Baseline (before intervention), 30 minutes after intervention, 2 hours after intervention, and prior to first mobilization (within 24 hours).
  Comfort level was assessed using the "General Comfort Scale Short Form" through face-to-face interviews at the same locations.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University Hospital, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No